CLINICAL TRIAL: NCT00811694
Title: Neurovascular Coupling in Patients With Open Angle Glaucoma
Status: Terminated | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjäger Mayrl, MD, Department of Clinical Pharmacology, Medical University of Vienna , Austria
Other Study IDs: OPHT-200104
Record Dates: First submitted 2008-07-02; First posted 2008-12-19 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Glaucoma
Keywords: glaucoma; ficker stimulation; ocular blood flow
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- a: 15 male and 15 female patients with glaucoma
  Interventions: Other: ocular blood flow measurements
- b: 30 sex matched healthy volunteers
  Interventions: Other: ocular blood flow measurements

INTERVENTIONS:
Other: ocular blood flow measurements — non-invasive haemodynamic measurements of retinal vessel diameters, laser Doppler flowmetry and laser Doppler velocimetry

SUMMARY:
A variety of studies demonstrate that ocular blood flow is altered in glaucoma. Various animal and human studies have shown an increase in retinal and optic nerve head blood flow in response to diffuse luminance flicker. Based on studies with ERG, this effect has been attributed to augmented activity in the retinal ganglion cells and associated axons indicating a coupling mechanism between neuronal activity and retinal blood flow. Whereas a variety of studies have confirmed these effects, the knowledge about this coupling in the retina of patients with glaucoma is sparse.

Recently the investigators could show that flicker induced vasodilatation is blunted in patients with open angle glaucoma. However, the investigators results are limited by the fact that only data about retinal vessel diameters, not blood flow per se, are available. The further development of the investigators current flicker stimulation technique now allows us to determine blood flow velocity during flicker stimulation. Thus, in the current study, the investigators set out to determine whether this blood flow response is impaired in patients with glaucoma as compared to those in healthy volunteers and whether this is related to altered neural activity.

The study objective was, to investigate whether the blood flow response to flicker stimulation is altered in patients with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 20 and 80 years.
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant.
* Inclusion criteria of patients are open angle glaucoma.
* Men and women will be included in equal parts. A pregnancy test will be performed at screening.
* Ametropia of less than 3 diopters and anisometropia of less than 1 diopter.

Exclusion Criteria:

* Treatment with vasoactive drugs.
* Presence of intraocular pathology other than open angle glaucoma.
* Presence of ocular hypertension or PEX (pseudoexfoliation) glaucoma
* History or family history of epilepsy.
* Pregnancy.
* Diabetes mellitus.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Retinal blood velocity (laser Doppler velocimetry) | measurements done only once on the studyday
Retinal arterial and venous diameter (Retinal vessel analyzer) | measurements done only once on the studyday
Optic nerve head blood flow (laser Doppler flowmetry) | measurements done only once on the studyday
Latency and amplitude (pattern ERG) | measurements done only once on the studyday

SECONDARY OUTCOMES:
Mean arterial pressure | measurements done only once on the studyday

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjäger Mayrl, MD, Principal Investigator — Department of Clinical Pharmacology, Meical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Meical University of Vienna, Austria, Vienna, Austria